CLINICAL TRIAL: NCT01083030
Title: Paclitaxel-coated Balloons in Femoral Indication to Defeat Restenosis
Acronym: PACIFIER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Saarland (Other)
Responsible Party: Sponsor
Organization: Universität des Saarlandes (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pac 12
Record Dates: First submitted 2010-03-04; First posted 2010-03-09 (Estimated); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Peripheral Artery Disease
Keywords: pAVK; PTA; drug coated balloon
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Angioplasty

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional PTA (Active Comparator): Angioplasty of SFA with uncoated balloon catheters
  Interventions: Device: Percutaneous transluminal angioplasty (PTA)
- Drug coated balloon (Experimental): Angioplasty of SFA with paclitaxel-coated balloon catheters
  Interventions: Combination Product: DCB

INTERVENTIONS:
Device: Percutaneous transluminal angioplasty (PTA) — Angioplasty of superficial femoral artery (SFA)
  Other Names: uncoated PTA
  Arms: Conventional PTA
Combination Product: DCB — Drug Coated Balloon Angioplasty
  Arms: Drug coated balloon

SUMMARY:
The aim of the study is correlating efficacy of the treatment to the proportion of paclitaxel-dose supplied by the catheter. Forty-five patients each will be treated by paclitaxel-coated or uncoated conventional balloon catheters in randomized order in 3 study centers. Main inclusion criteria are Rutherford class 2 - 5, ≥70% stenosis or occlusion in the superficial femoral or popliteal artery, main exclusion criteria are related to the use of paclitaxel and the need for follow-up examinations. Either clinical or angiographic follow-up examinations are planned 6, 12 and 24 months following the intervention. Primary endpoint is 6-month angiographic late lumen loss. Secondary endpoints are further angiographic and clinical efficacy and various safety criteria.

DETAILED DESCRIPTION:
Paclitaxel-coated balloons have been shown to reduce late lumen loss, restenosis rates and the need for repeat target lesion revascularization compared to conventional uncoated balloon catheters. The aim of the study is correlating efficacy of the treatment to the proportion of paclitaxel-dose supplied by the catheter. To this end paclitaxel loss of catheters in the introductory sheaths and residual paclitaxel on used balloons will be determined and correlated to individual data indicating inhibition of neointimal proliferation. According to the study protocol 45 patients each will be treated by paclitaxel-coated or uncoated conventional balloon catheters in randomized order in 3 study centers. Main inclusion criteria are Rutherford class 2 - 5, ≥70% stenosis or occlusion in the superficial femoral or popliteal artery, 3 to 30 cm of length; beyond common contraindications against PTA main exclusion criteria are related to the use of paclitaxel and the need for follow-up examinations. Patients will be blinded against treatment. Blinding of investigators after assignment of a patient to a treatment is not possible due to differences in the appearance of coated and uncoated catheters. Either clinical or angiographic follow-up examinations are planned 6, 12 and 24 months following the intervention. Primary endpoint is 6-month angiographic late lumen loss evaluated by a blinded independent core lab. Secondary endpoints are interventional success rate, restenosis rates, minimal lumen diameter, target lesion revascularization, change in Rutherford class, change in ankle-brachial-index, major amputations, a composite safety endpoint (defined as MAE =death of any cause, target limb amputation, clinically / DUS driven TLR) and all kinds of serious adverse events possibly related to the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with PAOD, Rutherford stage 2-5, Occlusion or stenosis >70% in diameter of at least 3 cm length in the superficial femoral artery and/ or popliteal artery

Exclusion Criteria:

* Acute thrombus or aneurysm in the index limb/ vessel
* Doubts in the willingness or capability of the patient to allow follow up examination

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2010-03; Primary Completion 2011-08 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Late lumen loss | 6 months
  Efficacy of paclitaxel coated percutaneous transluminal angioplasty (PTA) balloons in inhibiting restenosis of femoropopliteal arteries (late lumen loss)

SECONDARY OUTCOMES:
Angiographic and clinical efficacy measures | 6 months
  Various angiographic and clinical efficacy measures, safety and tolerance of paclitaxel coated PTA balloons in inhibiting restenosis of femoropopliteal arteries:
  1. Target lesion revascularization (Target lesion revascularization is defined as any reintervention or artery bypass graft surgery involving the target lesion.)
  2. Change in Rutherford stage compared to pretreatment
  3. Major amputations at the index limb
  4. Pre-defined event free survival

CONTACTS AND LOCATIONS:
Overall Officials: Michael Werk, MD, Principal Investigator — Martin-Luther-Hospital Berlin
Locations (3):
- Germany (3):
  - Vivantes - Klinikum Neukölln, Berlin
  - Ev. Hubertus Hospital Berlin, Berlin
  - Martin-Luther-Hospital Berlin, Berlin

REFERENCES:
- [Background] Scheller B, Hehrlein C, Bocksch W, Rutsch W, Haghi D, Dietz U, Bohm M, Speck U. Two year follow-up after treatment of coronary in-stent restenosis with a paclitaxel-coated balloon catheter. Clin Res Cardiol. 2008 Oct;97(10):773-81. doi: 10.1007/s00392-008-0682-5. Epub 2008 Jun 5. PMID 18536865
- [Background] Tepe G, Zeller T, Albrecht T, Heller S, Schwarzwalder U, Beregi JP, Claussen CD, Oldenburg A, Scheller B, Speck U. Local delivery of paclitaxel to inhibit restenosis during angioplasty of the leg. N Engl J Med. 2008 Feb 14;358(7):689-99. doi: 10.1056/NEJMoa0706356. PMID 18272892
- [Background] Scheller B, Hehrlein C, Bocksch W, Rutsch W, Haghi D, Dietz U, Bohm M, Speck U. Treatment of coronary in-stent restenosis with a paclitaxel-coated balloon catheter. N Engl J Med. 2006 Nov 16;355(20):2113-24. doi: 10.1056/NEJMoa061254. Epub 2006 Nov 13. PMID 17101615
- [Background] Scheller B, Speck U, Abramjuk C, Bernhardt U, Bohm M, Nickenig G. Paclitaxel balloon coating, a novel method for prevention and therapy of restenosis. Circulation. 2004 Aug 17;110(7):810-4. doi: 10.1161/01.CIR.0000138929.71660.E0. Epub 2004 Aug 9. PMID 15302790
- [Background] Werk M, Langner S, Reinkensmeier B, Boettcher HF, Tepe G, Dietz U, Hosten N, Hamm B, Speck U, Ricke J. Inhibition of restenosis in femoropopliteal arteries: paclitaxel-coated versus uncoated balloon: femoral paclitaxel randomized pilot trial. Circulation. 2008 Sep 23;118(13):1358-65. doi: 10.1161/CIRCULATIONAHA.107.735985. Epub 2008 Sep 8. PMID 18779447
- [Derived] Werk M, Albrecht T, Meyer DR, Ahmed MN, Behne A, Dietz U, Eschenbach G, Hartmann H, Lange C, Schnorr B, Stiepani H, Zoccai GB, Hanninen EL. Paclitaxel-coated balloons reduce restenosis after femoro-popliteal angioplasty: evidence from the randomized PACIFIER trial. Circ Cardiovasc Interv. 2012 Dec;5(6):831-40. doi: 10.1161/CIRCINTERVENTIONS.112.971630. Epub 2012 Nov 27. PMID 23192918